CLINICAL TRIAL: NCT05468658
Title: The Effect of Feng Shui Delivery Room Design on Maternal and Infant Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, ZULFIYYA NURALIYEVA, PhD, Assist. Prof. in Midwifery in Istinye University, Istinye University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IstanbulUC-1
Record Dates: First submitted 2022-03-10; First posted 2022-07-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Delivery Problem; Delivery Fear; Delivery; Injury; Birth; Prolonged; Birth Disorder
Keywords: Feng Shui; Birth; Philosophy; Midwifery care; Birth environment
MeSH Terms: conditions — Dystocia; Wounds and Injuries; Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (A): Feng Shui Birth Unit (Experimental): 1. The cabinets will be painted using salmon and pastel green.
  2. It is planned to make designs specific to the philosophy of Feng Shui on the doors and walls of the birthing unit.
  3. Live nature videos and sounds will be projected onto the wall.
  4. Fabric curtains will be replaced with curtains designed according to the philosophy of Feng Shui.
  5. Natural plants will be placed.
  6. Lighting will be used.
  7. Bed linen will be designed according to the Feng Shui.
  8. Wooden bell will be used.
  9. Turtle, elephant and Wu Lou objects will be placed.
  10. The Bagua mirror will be placed.
  11. Crystals will be placed.
  12. Natural stones will be placed.
  13. The fountain will be placed in the east compass direction of the unit.
  14. Straw bamboo separator will be used.
  Interventions: Other: Designing the birthing unit according to the philosophy of Feng Shui
- Control Group (B): Routine Birth Unit (No Intervention): The delivery unit of the institution consists of a small corridor, a labor room, a delivery room and a baby room. In the small corridor, there is a desk, document cabinets, vaccine cabinet and medicine cabinet for the midwife to work. The institution's routine delivery unit is equipped with standard medical devices and supplies. However, there are medical devices that are not used in the unit. White bed linens designed with the standard hospital logo are used in the unit. However, the curtains are plain cream, the walls are light blue, and the ceilings are white.

INTERVENTIONS:
Other: Designing the birthing unit according to the philosophy of Feng Shui — 1. The cabinets will be painted using salmon and pastel green.
  2. It is planned to make designs specific to the philosophy of Feng Shui on the doors and walls of the birthing unit.
  3. Live nature videos and sounds will be projected onto the wall.
  4. Fabric curtains will be replaced with curtains designed according to the philosophy of Feng Shui.
  5. Natural plants will be placed.
  6. Lighting will be used.
  7. Bed linen will be designed according to the Feng Shui.
  8. Wooden bell will be used.
  9. Turtle, elephant and Wu Lou objects will be placed.
  10. The Bagua mirror will be placed.
  11. Crystals will be placed.
  12. Natural stones will be placed.
  13. The fountain will be placed in the east compass direction of the unit.
  14. Straw bamboo separator will be used.
  Other Names: Unit design
  Arms: Experimental Group (A): Feng Shui Birth Unit

SUMMARY:
The aim of the study is to compare the births that took place in the Feng Shui Birth unit and those that took place in the standard delivery unit in terms of mother-infant health outcomes.

The study will be carried out in a private clinic in Istanbul, between July and December 2022. In the study, which is planned as a controlled experimental study, 50 women who applied first and met the inclusion criteria of the study will be selected as the Control Group (B), and it is planned that these women will give birth using the normal routine delivery unit of the clinic. It is planned that the next 50 women will form the Experimental Group (A): and give birth in the birth environment designed according to the Feng Shui Philosophy.

DETAILED DESCRIPTION:
This study is based on the hypothesis that the birth environment requires greater attention to ameliorate existing challenges in modern obstetric practice. The main focus is on the negative experiences that result from increased intervention during childbirth and the accompanying fear, anxiety, pain and stress. In order to reduce these emerging problems, it is planned to design the maternity unit based on the Feng Shui philosophy, inspired by the information obtained from the evidence-based health service design advocating bringing nature to the hospital.

Studies conducted abroad on what kind of birth environment women want and evidence-based guidelines. However, there is a need for such studies to be conducted in Turkey and for the creation of evidence-based guidelines by taking cultural characteristics into account. In line with this study, it is thought that planning and implementing new and positive birth environments with a multidisciplinary approach by architects, designers and health professionals will contribute positively to mother and baby health.

The dissemination of evidence-based good practices in obstetrics services to include all women giving birth is necessary in terms of the principle of quality service and equality. However, with this study, it is emphasized that the birth environment is not only limited to spatial arrangement, but is a matter of philosophy.

In this context, it is aimed to compare the births in the Feng Shui delivery unit with the ones that take place in the routine birth unit, with its design and decoration that will minimize the rate of anxiety, fear, pain, stress, emergency cesarean section, synthetic oxytocin and instrumental need, and increase the rates of maternal satisfaction and breastfeeding proficiency.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women;

* No Turkish communication problem,
* be at least 18 years old,
* No history of risky pregnancy
* Not having a chronic (Cardiovascular system diseases, Diabetes Mellitus, Hypertension, etc.) and mental (Major depression, Psychosis, etc.) disease,
* Having nulliparous pregnant women who will give birth to a singleton baby in the head delivery position,
* 37 to 42 weeks of gestational weeks of gestation,
* Pregnant women who are faced with cord entanglement, meconium amniotic fluid problems but decided to continue their vaginal delivery
* To be able to meet the criteria for saliva sampling, Having stopped eating at least 1.5 hours ago, Stopped consuming beverages containing caffeine in the last 2 hours, Not doing any strenuous physical activity in the last 1 hour, Not consuming alcohol within 24 hours, Not brushing teeth in the last 2 hours and no bleeding in the gums

Exclusion Criteria:

* Pregnant women who applied to the delivery unit between 21:00 and 06:00.
* Having a Body Mass Index (BMI) below 18.5 kg/m2 and above 24.9 kg/m2 during the pregnancy period,
* Newborn baby weighing less than 2.5 kg or over 4.5 kg,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Women's pain rates-before | Between 21:00 o'clock and 06:00 o'clock before birth
  H0= The women who give birth in a Feng Shui birthing unit will have lower pain rates than women who give birth in a routine birthing unit.
  H1= There is no difference between the rates of pain of a woman who gives birth in a Feng Shui delivery unit and the rates of pain a woman who gives birth in a routine delivery unit.
  The woman's pain, will be measured by the Visual Analog Scale (VAS). VAS is a symptom assessment tool where individuals mark on a horizontal/vertical bar that is 10 cm or 100mm. While the starting point of this tool shows no symptoms, the ending point shows the most severe state.
Women's stress rates-before | Between 21:00 o'clock and 06:00 o'clock before birth
  H0=The women who give birth in the Feng Shui delivery unit will have lower rates of stress than the women who give birth in the routine delivery unit.
  H1= There is no difference between the stress rates of a woman who gives birth in a Feng Shui delivery unit and tthe stress rates of a woman who gives birth in a routine delivery unit.
  The woman's stress will be measured with salivary cortisol kits. Cortisol assesment; İt is planned to look at cortisol values in order to express the stress level of women with objective data. Saliva samples will be taken from pregnant women to evaluate cortisol levels. Saliva samples will be collected through Salivette® (Sample Collection Tube, Sarstedt, Nümbrecht, Germany) brand saliva sample collection material.
Women's fear of childbirth rates | Between 21:00 o'clock and 06:00 o'clock before birth
  Ho=The women who give birth in the Feng Shui delivery unit will have lower rates of fear of childbirth than the women who give birth in the routine delivery unit.
  H1= There is no difference between the fear of childbirth rates of a woman who gives birth in a Feng Shui delivery unit and the fear of childbirth rates of a woman who gives birth in a routine delivery unit.
  Women's fear before childbirth will be measured by Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) version A scale.
  The W-DEQ version A is a 33-item scale. The answers in the scale are numbered from 0 to 5 and are in a six-point Likert type. A high item total score indicates a high level of fear.
  * W-DEQ score ≤ 37 mild,
  * W-DEQ score = 38-65 moderate,
  * W-DEQ score = 66-84 severe,
  * W-DEQ score ≥ 85 indicates clinical level of fear.
Women's fear of childbirth rates | 2 hours after birth
  H0=The women who give birth in the Feng Shui delivery unit will have lower rates of fear of childbirth than the women who give birth in the routine delivery unit.
  H1= There is no difference between the fear of childbirth rates of a woman who gives birth in a Feng Shui delivery unit and the fear of childbirth rates of a woman who gives birth in a routine delivery unit.
  Postpartum fears of women will be measured with Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) version B. In the measurement tool, there are a total of 33 questions including feelings and thoughts such as fear, confidence, feeling of loneliness, and happiness.
  The scale is one-dimensional. Scores from the scale range from 33 to 198. If the scores obtained from the scale are lower than 37, it means low-grade fear of childbirth, between 38-65 indicates moderate fear of childbirth, 66-84 indicates severe fear of childbirth, and above 85 indicates clinical-grade fear of childbirth (Uçar, 2013).
Labor time | between 10-15 hours on average
  H0=The labor period of the woman who give birth in the Feng Shui delivery unit will have shorter than the woman who give birth in the routine delivery unit.
  H1= There is no difference between the labor period of a woman who gives birth in a Feng Shui delivery unit and the labor period a woman who gives birth in a routine delivery unit.
The intervention (use of synthetic oxytocin, use of instrumental, resorting to episiotomy, urgent need for cesarean section) | between 10-15 hours on average
  H0= The rate of intervention to women in the Feng Shui delivery unit will have lower than the rate of intervention to women in the routine delivery unit (use of synthetic oxytocin, use of instrumental, resorting to episiotomy, urgent need for cesarean section).
  H1= There is no difference between the rates of intervention of a woman who gives birth in a Feng Shui delivery unit and the rates of intervention a woman who gives birth in a routine delivery unit.
Women's concern rates-before | Between 21:00 o'clock and 06:00 o'clock before birth
  H0=The women who give birth in the Feng Shui delivery unit will have lower rates of concern than the women who give birth in the routine delivery unit.
  H1= There is no difference between the rates of concern of a woman who gives birth in a Feng Shui delivery unit and the rates of concern a woman who gives birth in a routine delivery unit.
  The woman's concern will be measured by the Visual Analog Scale (VAS). VAS is a symptom assessment tool where individuals mark on a horizontal/vertical bar that is 10 cm or 100mm. While the starting point of this tool shows no symptoms, the ending point shows the most severe state.
Women's concern rates-after | 2 hours after birth
  H0=The women who give birth in the Feng Shui delivery unit will have lower rates of concern than the women who give birth in the routine delivery unit.
  H1= There is no difference between the rates of concern of a woman who gives birth in a Feng Shui delivery unit and the rates of concern a woman who gives birth in a routine delivery unit.
  The woman's concern will be measured by the Visual Analog Scale (VAS). VAS is a symptom assessment tool where individuals mark on a horizontal/vertical bar that is 10 cm or 100mm. While the starting point of this tool shows no symptoms, the ending point shows the most severe state.
Women's pain rates-after | 2 hours after birth
  H0= The women who give birth in the Feng Shui delivery unit will have lower rates of pain than the women who give birth in the routine delivery unit.
  H1= There is no difference between the rates of pain of a woman who gives birth in a Feng Shui delivery unit and the rates of pain a woman who gives birth in a routine delivery unit.
  The woman's pain, will be measured by the Visual Analog Scale (VAS). VAS is a symptom assessment tool where individuals mark on a horizontal/vertical bar that is 10 cm or 100mm. While the starting point of this tool shows no symptoms, the ending point shows the most severe state.
Women's stress rates-after | 2 hours after birth
  The women who give birth in the Feng Shui delivery unit will have lower rates of stress than the women who give birth in the routine delivery unit.
  The woman's stress will be measured with salivary cortisol kits. Cortisol assessment; İt is planned to look at cortisol values in order to express the stress level of women with objective data. Saliva samples will be taken from pregnant women to evaluate cortisol levels. Saliva samples will be collected through Salivette® (Sample Collection Tube, Sarstedt, Nümbrecht, Germany) brand saliva sample collection material.

SECONDARY OUTCOMES:
The satisfaction | 2 hours after birth
  H0=The satisfaction rate of the woman who give birth in the Feng Shui delivery unit will higher than the woman who give birth in the routine delivery unit.
  H1= There is no difference between the the satisfaction rate of a woman who gives birth in a Feng Shui delivery unit and the satisfaction rate the a woman who gives birth in a routine delivery unit.
  Birth satisfaction of women at stage 4 of labor will be measured with the Birth Satisfaction Scale-Revised (BSS-R).
  The scale consists of 10 items and 3 sub-dimensions. The total raw score ranges from 0-40. As the total score obtained from the scale increases, the satisfaction level of women with the care they receive at the hospital increases. In this study, scale cut-off scores were calculated by dividing the total score into three equal parts: - (1) low satisfaction <13 points, (2) moderate satisfaction 14-27 points, (3) high satisfaction ≥28 points.
Breastfeeding proficiency rate | 2 hours after birth
  H0=The postpartum breastfeeding adequacy ratio scores will higher for a woman who gives birth in a Feng Shui delivery unit compare to a woman who gives birth in a routine delivery unit.
  H1= There is no difference between the breastfeeding proficiency rate of a woman who gives birth in a Feng Shui delivery unit and breastfeeding proficiency rate the a woman who gives birth in a routine delivery unit.
  Breastfeeding proficiency rate will be measured with the Bristol Breastfeeding Scale. The tool was developed to measure frequently encountered postpartum breastfeeding difficulties and its validity has been approved.
  The scale is a Likert-type scale comprising the 4 items of "positioning," "holding," "sucking" and "swallowing." Each item is scored between 0- 2 points. The lowest possible score on the scale is 0, the highest is 8. Lower scores indicate that the breastfeeding is not successful, the higher scores signify successful breastfeeding.
Breastfeeding initiation time | one minute after birth
  H0=Breastfeeding initiation time will shorter for a woman who give birth in a Feng Shui delivery unit compare to a woman who give birth in a routine delivery unit.
  H1= There is no difference between the breastfeeding initiation time of a woman who gives birth in a Feng Shui delivery unit and breastfeeding initiation time the a woman who gives birth in a routine delivery unit.
APGAR score | one minute after birth
  H0=APGAR scores will higher for a woman who give birth in a Feng Shui delivery unit compare to a woman who give birth in a routine delivery unit.
  H1= There is no difference between the APGAR scores of a woman who gave birth in a Feng Shui delivery unit and the APGAR scores of a woman who gave birth in a routine delivery unit.

CONTACTS AND LOCATIONS:
Overall Officials: ZULFIYYA NURALIYEVA, PhD, Study Director — Istinye University; GULUMSER DOLGUN, PHD, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Private Mediplus Medical Center, Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No